CLINICAL TRIAL: NCT05838885
Title: A Multicenter, Randomized, Open-label, Positive-controlled Phase 2 Study to Explore the Optimal Dose of Y- Shaped Pegylated Recombinant Growth Hormone (YPEG-rhGH) in Children With Short Stature (ISS, SGA, TS)
Brief Title: A Trial of YPEG-rhGH in Children With Short Stature
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB2106GH
Record Dates: First submitted 2023-03-21; First posted 2023-05-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Short Stature; Small for Gestational Age; Turner Syndrome
Keywords: Growth hormone; Somatotropin; Short stature; Idiopathic short stature; Small for gestational age; Turner syndrome
MeSH Terms: conditions — Turner Syndrome; Dwarfism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YPEG-GH low dose group (Experimental)
  Interventions: Drug: YPEG-rhGH
- YPEG-GH high dose group (Experimental)
  Interventions: Drug: YPEG-rhGH
- rhGH low dose group (Active Comparator)
  Interventions: Drug: rhGH
- rhGH high dose group (Active Comparator)
  Interventions: Drug: rhGH

INTERVENTIONS:
Drug: YPEG-rhGH — YPEG-rhGH, 140μg/kg, s.c., once a week, for 52 weeks
  Arms: YPEG-GH low dose group
Drug: YPEG-rhGH — YPEG-rhGH, 280μg/kg, s.c., once a week, for 52 weeks
  Arms: YPEG-GH high dose group
Drug: rhGH — rhGH, 245μg/kg/week, divided into 7 subcutaneous injections, once daily, for 52 weeks
  Arms: rhGH low dose group
Drug: rhGH — rhGH, 470μg/kg/week, divided into 7 subcutaneous injections, once daily, for 52 weeks
  Arms: rhGH high dose group

SUMMARY:
To explore the dose-response relationship between pharmacokinetics and pharmacodynamics of Y- Shaped Pegylated growth hormone injection (YPEG-GH) in children with short stature (idiopathic short stature (ISS), small for gestational age (SGA), Turner syndrome (TS)).

To evaluate its tolerability, safety and efficacy and to provide evidence for dose selection and titration for future clinical development and clinical application in these population.

ELIGIBILITY:
Inclusion Criteria:

1. Prepubertal (Tanner I), aged older than 4 years and younger than10 years for girls and 11 years for boys.
2. Body weight: 12kg ≤ body weight ≤ 50kg.
3. For children with idiopathic short stature: a) Birth length and weight were at the 10th percentile and above of normal reference values for infants of the same gestational age and sex; b) Height at screening was 2.0 standard deviations (SD) below the mean height for chronological age and sex c) Exclude other causes such as systemic diseases, other endocrine diseases, nutritional diseases, chromosomal abnormalities, skeletal dysplasia, psycho-emotional disorders, etc. were excluded d) GH peak ≥10.0ng/ml confirmed by two different drug GH provocation tests; e) Bone age (BA)-chronological age (CA) ≤1 year.
4. For children with small for gestational age: a) Birth length and weight were at the 10th percentile and below the normal reference values for infants if the same gestational age and sex; b) Gestational age at birth ≥ 24 weeks; c) Height at screening was below -2 SD of the mean for the same age and sex, and please refer to the protocol annex 1 for height.
5. For children with Turner syndrome: a) Chromosome karyotype: 45, X; 45, X/46, XXqi; 45, X/46, XXr; 45, X/46, XX; 46, XXqi; 46, XXpi; 45, X/47, XXX; 46, XXp-; 45, X/46, XXp-; 46, XXq-; 45, x/46, XXq-; 45, X/46, XX/47, XXX, etc.; b) Having at least one specific physical characteristic: Including but not limited to low posterior hairline, facial skin nevus, neck flips, short neck, low ear position, small jaw, high palatal arch, shield chest, wide breast spacing, elbow ectropion, knee ectropion, short 4th and 5th metacarpal, nail dysplasia, scoliosis, ptosis, strabismus, cardiovascular system abnormalities such as aortic stenosis, bicuspid aortic valve, hypertension, and reproductive system abnormalities such as primary gonadal insufficiency, renal malformation, hypothyroidism and middle ear disease; c) The height at screening was below the mean -2SD of the same age and gender, and please refer to the protocol annex 1 for height.
6. Understands and signs the informed consent form voluntarily by the subject's parent(s) and/or legal guardian(s). And written assent of the subject is required if the subject is 8 years of age or older).

Exclusion Criteria:

1. For children with small for gestational: confirmed or suspected Bloom syndrome.
2. For children with Turner syndrome: containing a Y chromosome or a fragment derived from a Y chromosome.
3. Children with closed epiphysis.
4. Children who diagnosed or highly suspected growth hormone deficiency (GHD), or other types of growth abnormalities: e.g., Noonan syndrome, Prader-Willi syndrome, Russell-Silver syndrome, etc.
5. Children who have previously received systemic growth-promoting therapy, including but not limited to rhGH, aromatase inhibitors, sex hormones, etc., for at least 1 month or longer.
6. Children who are now receiving or plan to receive the therapy of glucocorticoids, methylphenidate, and any other drugs that may have an effect on growth.
7. Children with abnormal values of liver and kidney function (ALT > 1.5 ULN, Cr > 1 ULN).
8. Concomitant with chronic hepatitis B, AIDS, tuberculosis, and any other chronic infectious disease.
9. Patients with severe allergic constitutions or allergic to growth hormone or its excipients such as mannitol, lysine, sodium chloride and other ingredients.
10. Patients with a previous history of malignancy or are currently suffering from active malignancy, including intracranial tumors.
11. Patients with abnormal glucose regulation (including abnormal fasting glucose and/or abnormal glucose tolerance) or diabetes.
12. Patients who are mentally ill or have a family history of mental illness.
13. Patients who are suffering from chronic systemic diseases, such as malnutrition, immunocompromised individuals, asthma, etc.
14. Patients with congenital intracranial hypertension.
15. Patients with slipped capital femoral epiphysis (SCFE).
16. Patients with scoliosis exceeding 15°;
17. Patients who have participated in any drug clinical study (as a subject) within 3 months prior to screening and have received a drug intervention
18. Patients who the investigators considered unfit for the study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic-area under plasma concentration versus time curve | up to 52 weeks
Pharmacokinetic-maximum serum concentration | up to 52weeks
Pharmacokinetic-time to reach the maximum plasma concentration | up to 52 weeks
Pharmacokinetic-terminal disposition phase half-life | up to 52 weeks
Pharmacokinetic-terminal elimination rate constant | up to 52 weeks
Pharmacokinetic-apparent clearance after extravascular administration | up to 52 weeks
Pharmacokinetic-apparent volume of distribution | up to 52 weeks

SECONDARY OUTCOMES:
Pharmacodynamics-the properties of Insulin-like growth facto1 and Insulin-like growth factor binding receptor 3. | up to 57 weeks
Height velocity (HV, cm/year) | At 52 weeks of treatment
Change of height velocity compared to baseline (ΔHV, cm/year) | At 52 weeks of treatment
Height standard deviation according to chronological age (Ht SDS CA) | At 52 weeks of treatment
Change in bone age | At 52 weeks of treatment
Adverse events (including injection site reactions), changes from baseline in vital signs and laboratory tests | up to 57 weeks

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The Fourth Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sanya Central Hospital (Hainan Third People's Hospital), Sanya, Hainan
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Children's Hospital, Capital Institute of Pediatrics, Beijing
  - Children's Hospital of Shanghai, Shanghai